CLINICAL TRIAL: NCT06406036
Title: Reliability and Validity of Rivermead Mobility Index in Urdu Language Among Pakistani Stroke Population
Brief Title: A Validity and Reliability Study for Urdu Version of Rivermead Mobility Index in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0293
Record Dates: First submitted 2022-06-27; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Rivermead Mobility Index; Urdu Version; Reliability; Validity; Stroke; Mobility
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to translate and cross-culturally adapt the Rivermead mobility index questionnaire into traditional Urdu language to investigate its psychometric properties (reliability & validity) for those patients who are confronting stroke.

DETAILED DESCRIPTION:
As per preceding commendation, Rivermead Mobility Index will be translated into Urdu language from its English version and adapted culturally in Pakistan. Among Stroke population, Rivermead Mobility Index will be conducted in 50 patients recruited by convenience sampling technique under the pre-defined inclusion and exclusion criteria after signing consents forms. For testing inter-observer reliability and intra-observer reliability of Rivermead Mobility Index, Barthel Index and Functional Independence Measure will be administrated by two observers, on the same day, with a time interval of 2 hours between 1st and 2nd conduction. As for the 3rd conduction, it will be carried out after seven days by the first observer, for intra-observer assessment. Statistical Package of Social Sciences software version 24 has been used for the purpose of data entry and analysis. Internal consistency will be assessed by using an intra-class correlation coefficient. The Rivermead Mobility Index will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female both genders
* Adults between the ages of 18 and above
* Stroke patients ( chronic)
* Ability to provide informed consent

Exclusion Criteria:

* Any musculoskeletal pathologies
* Suffering from any cardiovascular pathologies
* Any history of fracture
* Any histories of infections
* Any history of neurological disorders
* Having any spinal deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population for this study will be diagnosed cases of stroke.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Rivermead Mobility Index | 1st day
  The Rivermead Mobility index is a standardized assessment tool to investigate patients work and activity specific physical disability related to work. Rivermead Mobility Index scale have 15 items.
Barthel Index | 1st day
  The Barthel Index is an ordinal scale that is used to assess performance in daily activities. A higher number reflects better capacity to operate independently upon hospital release.
Functional Independence Measure | 1st day
  Functional Independence Measure instrument was designed for assessing responsive changes throughout the course of a complete inpatient medical rehabilitation programme. The instrument is used to determine a patient's level of impairment as well as any changes in their condition as a result of rehabilitation or medical treatment. Is an 18-item, seven-level, ordinal scale intended to be sensitive to changes over the course of a comprehensive inpatient medical rehabilitation program.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No